CLINICAL TRIAL: NCT04362488
Title: Evaluation of Ankle Propriocement and Stability in Patients Affected by Traumatic Lateral Ankle Instability Before and After External Ankle Ligament Recontruction
Brief Title: Evaluation of Ankle Propriocement and Stability
Acronym: ANKLE-INT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 558/2018/Oss/IOR
Record Dates: First submitted 2019-02-08; First posted 2020-04-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Ankle Sprains; Instability, Joint
Keywords: sprain; Brostrom; ankle instability
MeSH Terms: conditions — Ankle Injuries; Joint Instability; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: All patients who undergo surgery for a ankle lateral ligament reconstruction from 4th Febbruary 2019 till to the end of the study on 4th August 2020
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic post-traumatic lateral ankle instability (Experimental): The study population consists in patients affected by chronic post-traumatic lateral ankle instability who must undergo surgical intervention of ankle external ligament reconstruction.
  The patients will be analyzed pre and postoperatively using differents tests, questionnaires, instrument and clinical evaluation:
  * Delos system (computerized oscillating platform)
  * Foot and Ankle Ability Measure (FAAM), l'American Orthopaedic Foot and Ankle Score (AOFAs), SF12 questionnaires
  * modified Star Excursional Balance Test (mSEBT) and Short Physical Performance Battery (SPPB)
  Interventions: Procedure: Preoperative evaluation; Procedure: Postoperative evaluation

INTERVENTIONS:
Procedure: Preoperative evaluation — Preoperative evaluation using differents clinical evaluation tests, questionnaires, and instrument:
  * Delos system (computerized oscillating platform)
  * Foot and Ankle Ability Measure (FAAM), l'American Orthopaedic Foot and Ankle Score (AOFAs), SF12 questionnaires
  * modified Star Excursional Balance Test (mSEBT) and Short Physical Performance Battery (SPPB)
  Other Names: Questionnaires: "FAAM", "AOFAs", "SF12"; Instrument: "Delos computerized oscillating platform"; Tests: "mSEBT", "SPPB"
Procedure: Postoperative evaluation — Postoperative evaluation at 4 months of follow up after surgery using differents clinical evaluation tests, questionnaires, and instrument:
  * Delos system (computerized oscillating platform)
  * Foot and Ankle Ability Measure (FAAM), l'American Orthopaedic Foot and Ankle Score (AOFAs), SF12 questionnaires
  * modified Star Excursional Balance Test (mSEBT) and Short Physical Performance Battery (SPPB)
  Other Names: Questionnaires: "FAAM", "AOFAs", "SF12"; Instrument: "Delos computerized oscillating platform"; Tests: "mSEBT", "SPPB"

SUMMARY:
The objective of the study is to evaluate the postural control and proprioception before and after external capsulo-ligament reconstruction for ankle instability.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the postural control and proprioception before and after external capsulo-ligament reconstruction for ankle instability using differents tests, questionnaires and instrument:

* Delos system (computerized oscillating platform)
* Foot and Ankle Ability Measure (FAAM), l'American Orthopaedic Foot and Ankle Score (AOFAs), SF12 questionnaires
* modified Star Excursional Balance Test (mSEBT) and Short Physical Performance Battery (SPPB)

ELIGIBILITY:
Inclusion Criteria:

* patients who must undergo surgery;
* patients of both sexes aged between 18-40 years;
* patients who have given their informed written consent to participate in the study;
* patients who have given their consent to reach the Hospital to perform the 4-month check-up

Exclusion Criteria:

* patients with BMI> 30 kg / m2;
* patients with rheumatoid arthritis;
* patients with chronic inflammatory joint diseases;
* patients with pre-existing abnormalities of the ambulatory kinematics (amputations, neuro-muscular diseases, polio, hip dysplasias);
* patients with Severe arthrosis of the ankle (Kellgren-Lawrence> 3);
* patients with Severe knee arthritis (Kellgren-Lawrence> 3);
* patients with ACL injury;
* patients with severe postural instability;
* patients with cognitive impairments;
* patients with concomitant neurological diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Delos (computerized oscillating platform) | End of the study, 18 month from the beginning (04 August 2020)
  The patients will be analyzed pre and postoperatively using a computerized oscillating platform that shows the response of the foot as an adaptation to the ground. The result is expressed through stability index (%) compared to the average of the population.
Foot & Ankle Ability Measure (FAAM) questionnaire. | End of the study, 18 month from the beginning (04 August 2020)
  FAAM: expresses the personal evaluation of the patient on his difficulty in performing activities using 5 values for each question: no difficulty, slight difficulty, moderate difficulty, extreme difficulty, inability.
American Orthopaedic Foot & Ankle score (AOFAs) questionnaire | End of the study, 18 month from the beginning (04 August 2020)
  AOFAs: values from 0 to 100 dependent on limitations in performing activities
Short Form Health Survey - 12 questionnaire | End of the study, 18 month from the beginning (04 August 2020)
  SF12: personal assessment of one's state of health using multiple-answer questions with different values for each question.
modified Star Excursional Balance Test (mSEBT) functional test | End of the study, 18 month from the beginning (04 August 2020)
  mSEBT: best value resulting from the 3 equilibrium tests standardized for the length of the limb. The tests consist in reaching the greater distance with a foot along three (inverted Y-shaped) axes with between them an angle of 90 ° (rear) and two of 135 ° (antero-medial and anterior-lateral) while the opposite foot remains still on the ground
Short Physical Performance Battery functional test | End of the study, 18 month from the beginning (04 August 2020)
  The SPPB scale is a short battery of tests designed to evaluate the functionality of the lower limbs. This battery consists of 3 different sections. The total score of the scale has a range from 0 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Mosca, Principal Investigator — Rizzoli Orthopaedic Istitute, Bologna
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04362488/Prot_SAP_000.pdf